CLINICAL TRIAL: NCT06586996
Title: The Construction of Bidirectional Column Study and Prognosis Prediction of Acute Osteoporotic Vertebral Compression Fractures Based on Imaging and Clinical Data
Brief Title: The Construction of Bidirectional Column Study of Acute Osteoporotic Vertebral Compression Fractures
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: M2021606
Record Dates: First submitted 2024-09-04; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-01

CONDITIONS: Osteoporosis Fracture
Keywords: osteoporosis fracture
MeSH Terms: conditions — Osteoporotic Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- osteoporotic vertebral compression fractures
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
Our research group plans to establish a disease specific bidirectional cohort study on prognosis prediction of acute osteoporotic vertebral compression fracture based on imaging and clinical data, and to establish a comprehensive bioinformation database on OVCFs, including patient status, clinical data, laboratory examination, and imaging examination database

ELIGIBILITY:
Inclusion Criteria: all patients who suffer a acute osteoporosis vertebral compression fractures -

Exclusion Criteria: those who have endocrine disease which have impacts on the bone density

-

Ages: 50 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All the acute osteoporosis vertebral compression fracture patients who search for treatments in our hospital
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
VAS value | 2 weeks, 1 month, 2 months, 3months, 6 months and 12 months
  the visual analogue scale value of patient
vertebrae height | 2 weeks, 1 month, 2 months, 3months, 6 months and 12 months
  the height of the vertebrae according to the X rays
T value | 6months and 12 months
  the T value of the dual energy X-ray absorptiometry

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Third Hospita, Beijing, China